CLINICAL TRIAL: NCT06514937
Title: Efficacy of the E-motional Training Program for Improving Social Cognition in People With Dual Pathology in a Clinical and Prison Environment: Neuropsychological and Proteomic Study
Brief Title: Efficacy of the E-motional Training Program for Improving Social Cognition in People With Dual Pathology in a Clinical and Prison Environment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacin Biomedica Galicia Sur (Other)
Collaborators: Plan Nacional sobre Drogas (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023I086
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Social Behavior
Keywords: dual pathology
MeSH Terms: conditions — Social Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with dual pathology without social cognition damage (No Intervention): Patients with dual pathology without damage without intervention
- Patients with dual pathology with Social Cognition damage control (No Intervention): Patients with dual pathology with social cognition damage with regular therapy in the centre
- Patients with dual pathology with social cognition with Emotional Training (Experimental): Patients with dual pathology with social cognition damage with Emotional Training therapy in the centre
  Interventions: Behavioral: Emotional Training

INTERVENTIONS:
Behavioral: Emotional Training — Emotional Training Therapy following the programme in the computer
  Arms: Patients with dual pathology with social cognition with Emotional Training

SUMMARY:
Drug use, substance-related disorders (SUD), other addictive behaviors, or, from a broader perspective, dual pathology, are problems of enormous socio-health impact that still require a great research effort to improve diagnostic and therapeutic procedures employed in healthcare practice.

Since addictive behaviors have been consistently associated with the presence of alterations in cognitive and executive functions, it is necessary to be able to detect, evaluate, and have specific therapies for these dysfunctions and investigate, among other issues, the role they play in the onset and course of evolution. After implementing neuropsychological evaluation techniques for diagnostic improvement, the search addresses procedures that allow working on cognitive and executive deficits as a specific therapeutic target.

In a previous project, the investigators studied the presence of social cognition (SC) dysfunctions in a clinical sample of patients treated in drug addiction care facilities. The investigators evaluated the therapeutic efficacy of the ET® program in those who presented difficulties in SC and analyzed molecular patterns in saliva that could be associated with SC dysfunctions and predict therapeutic response. The ET® program is an online self-training program for SC rehabilitation that includes modules for emotion recognition (ER), Theory of Mind (ToM), and attributional style (AS).

To replicate the RCT carried out in patients with SUD in patients with dual pathology with difficulties in ER or ToM, in addition to including a gender perspective, tele-neuropsychology, and searching for a biomarker or a pattern of them that predicts the patient profile that will benefit from the training, using advanced LC-ESI proteomics techniques. It is also intended to subsequently improve the instrument (ET®) through the implementation of a gender perspective and big data analysis and machine learning, and the introduction of automated user management.

From the perspective of the STATE PLAN FOR SCIENTIFIC AND TECHNICAL RESEARCH AND INNOVATION, the project combines clinical and translational research, based on evidence of scientific and technological knowledge, and the use of e-health enabling technologies in the area of Health Services. Health for people with dual pathology, with special attention to the gender perspective.

DETAILED DESCRIPTION:
HYPOTHESIS There is evidence of the existence of social cognition (SC) dysfunctions in patients with SUD, and its potential implications in the etiopathogenesis, clinical course, and response to treatment have been postulated. At the healthcare level, SC should be taken into account in diagnostic and therapeutic procedures.

The detection of SC dysfunctions and the implementation of specific treatment for them will contribute to improving the therapeutic response of patients with SUD.

The general hypotheses of the study will be:

1. A high percentage of people with dual pathology and impairment of social cognition will be detected.
2. People with dual pathology and impairment of social cognition will improve after the intervention with the updated version of ET®.
3. A panel of potential biomarkers that predict therapeutic response can be identified.

GENERAL OBJECTIVES:

1. Determine the prevalence of dual pathology in clinical and prison samples of people with SUD.
2. Evaluate the presence of alterations in the domains that make up social cognition (SC) in people with dual pathology in clinical and prison samples.
3. Check the effectiveness of a computerized rehabilitation program for SC, the ET® program, in people with dual pathology who present SC dysfunctions.
4. Develop a panel of biomarkers in saliva that predicts which people with dual pathology will benefit from training, using shotgun mass spectrometry techniques (LC-ESI-MS/MS).
5. Conduct the study taking into account the gender perspective.

SPECIFIC OBJECTIVES:

1.1 Assess the prevalence of mental disorders in people with an addictive disorder.

1.2 Evaluate the differences in clinical and penitentiary environments of mental disorders in people with an addictive disorder.

1.3 Assess sex differences in the prevalence of mental disorders in people with an addictive disorder.

2.1 Evaluate the presence of dysfunctions in the SC of people with dual pathology.

2.2 Evaluate the dysfunctions in the subdomains of SC of people with dual pathology.

2.3 Evaluate the differences in clinical and penitentiary environments in SC dysfunctions in dual pathology.

2.4 Evaluate sex differences in SC dysfunctions in dual pathology.

3.1 Evaluate the effectiveness of the new version of the ET® program in people with dual pathology.

3.2 Evaluate the effectiveness of the new version of the ET® program on therapeutic response: adherence, quality of life, symptom perception, and relapses.

3.3 Evaluate the differences in clinical and prison settings in the effectiveness of treatment with ET®.

3.4 Assess gender differences in the efficacy of ET® treatment.

4.1 Increase the bank of saliva samples for proteomic studies. 4.2 Identify molecular patterns in saliva that are associated with SC dysfunctions.

4.3 Identify biomarkers that predict therapeutic response. 4.4 Evaluate gender differences in the study of biomarkers.

Methodology (subjects, variables, data collection, analysis plan):

To study the presence of SC dysfunctions in a clinical sample of patients treated in drug addiction care facilities, patients with a diagnosis of SUD who begin treatment in care centers in Galicia, Madrid, and Portugal, and in the prison in Cuenca will be recruited to carry out the phase of collecting sociodemographic variables, descriptive data, and psychometric evaluation using the battery described below.

To study the therapeutic efficacy of the ET® program in patients with dual pathology who present SC dysfunctions, a multicenter, longitudinal, prospective, controlled, and randomized multimodal (proteomic, neurocognitive, and clinical) study phase on the effectiveness of ET® will be carried out. Early prediction of response in patients with dual pathology requiring social cognition rehabilitation treatment. The response will be evaluated after 3 months (short term), after 12 sessions where activities on emotions and theory of mind are combined, and a follow-up will be carried out after 12 months (long term).

To identify new biomarkers in saliva, using mass spectrometry techniques (LC-ESI-MS/MS), which contribute to predicting which patients would benefit from receiving therapy with the ET® program, saliva samples will be collected to carry out the proteomic study in all participants in the ET® efficacy trial. To improve the ET® instrument to serve new types of users, both in healthcare and educational environments, and for its future adaptation for commercial exploitation, observations and evaluations of researchers and patients will be recorded to implement potential future ET® improvements.

STUDY POPULATION:

Patients who begin treatment in care facilities of the drug addiction network and prison, who meet the selection criteria specified in the inclusion criteria section and who do not meet any of the exclusion criteria.

NEUROPSYCHOLOGICAL ASSESSMENT (pre and post):

The neuropsychological evaluation time is estimated at 120 minutes. For the proposed protocol, at least 2 evaluation sessions are required:

* The assessment of dual pathology requires a 30-minute session.
* The assessment of social cognition requires 1 session of 30 minutes and 1 session of 60 minutes.

Patients will be evaluated before and after the intervention, and the evaluation will be repeated after 12 months, using the instruments described below:

Clinical evaluation:

* Dual Pathology Screening Interview (ECDD)
* Symptom Checklist-90-R (SCL-90-R)

Assessment of Social Cognition:

* The Interpersonal Reactivity Index (IRI)
* Ekman 60 Faces Test
* Movie for the Assessment of Social Cognition (MASC)
* Marlowe-Crowne Social Desirability Scale (MCSDS)
* Ambiguous Intentions Hostility Questionnaire (AIHQ)

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with dual pathology according to DSM-5 diagnosed by an expert clinician.
* Have the capacity to consent (competence).
* Read the project information sheet and sign the informed consent.
* Age>18 years-old

Exclusion Criteria:

* Illiterate
* History of moderate or severe neurological pathology (TBI, stroke, etc.),
* Current acute psychiatric process
* Abstinence of less than 15 days,
* Advanced cognitive impairment that does not allow evaluation.
* Have participated in another similar study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The participant eligibility is based of gender identity
Enrollment: 250 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Assess the presence of dysfunctions in the subdomains of social cognition | up to 12 months
  Social cognition by Ekman 60 Faces Test minimum and maximum values: 0 - 60 higher scores mean a better outcome.

SECONDARY OUTCOMES:
Accuracy and efficacy of ET® in patients with dual pathology | up to 12 months
  Social cognition by Movie for Assessment Social Cognition (MASC) minimum and maximum values: 0 - 51 higher scores mean a better outcome.

IPD SHARING:
Plan to Share IPD: No